CLINICAL TRIAL: NCT01324674
Title: Relationship Between Treatment With Bach´s Flower Remedy and Spiritual Well-Being of People With Common Mental Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: University of Sao Paulo (Other); Universidade do Vale do Paraíba (Other)
Responsible Party: Principal Investigator, Ana Paula Corrêa Castello Branco Nappi Arruda, MSc, Doctoral degree, UPECLIN HC FM Botucatu Unesp
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: upeclin/HC/FMB-Unesp-50
Record Dates: First submitted 2011-02-21; First posted 2011-03-29 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2011-03

CONDITIONS: Mental Disorders; Personal Well Being
Keywords: Common Mental Disorder; Efficacy of Bach´s flower remedy; Spiritual well-being
MeSH Terms: conditions — Mental Disorders | interventions — Complementary Therapies; Flower Essences

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo group (Placebo Comparator): Is the group of subjects that will take placebo
  Interventions: Other: Placebo group
- experimental group (Experimental): Is the group of subjects that will take Bach´s Flower remedies
  Interventions: Other: Bach´s Flower Remedy

INTERVENTIONS:
Other: Bach´s Flower Remedy — The subjects will have 4 drops 4 times per day, for approximately 8 months.
  Other Names: Complementary Alternative Therapy; Flower remedy
  Arms: experimental group
Other: Placebo group — The subjects will have a solution non-drug type, 4 drops 4 times per day, for approximately 8 months
  Other Names: Complementary Alternative Therapy
  Arms: Placebo group

SUMMARY:
The Common Mental Disorders (CMD) refer to health states involving non-psychotic psychiatric symptoms. Part of this broad diagnostic category, symptoms such as difficulty concentrating, forgetfulness, insomnia, fatigue, irritability, feelings of worthlessness, somatic complaints, etc. The CMD has a big social impact, and its prevalence in the general population is 25% and graduate students in health care reaches 40%. The Bach´s Flower Remedies are considered a complementary therapy approved and recommended by World Health Organization and by the Brazilian Ministry of Health and in his theory it has great spiritual nature. In addition, international scientific research have suggested that the strengthening of spiritual well-being can help significantly and positively promoting mental health. This project aims to assess the relationship between treatment with Bach´s Flower Remedies and Spiritual well-being of people with Common Mental Disorders in undergraduate health students of a university located in São José dos Campos, state of São Paulo, Brazil. This research presents a quantitative and qualitative methodology, experimental clinical trial, triple blind. The treatment will take place with two groups of forty people, the group of treatment and the placebo´s. The trial will happen in six sessions at intervals of 30 days, totaling eight months of treatment. Statistical analysis will be used chi-square or Fisher exact test to study the association between the scale of spiritual well-being and the use of Bach Flowers for each time point (3 times). To compare the evolution of the results (scales) during the study will set a model for ordinal data with repeated measurements over time. For these statistical tests is assumed a significance level of 5% (p < 0.005).

ELIGIBILITY:
Inclusion Criteria:

* People over 18 years old
* People who have read and agreed to participate by signing an informed consent
* People who obtain scores equal to or above 8 for women and equal to or above 6 for men in SRQ - 20
* People who does not ingest medication
* People who does not use any type of complementary therapy and integrative such as Herbal Medicine, Aromatherapy, Homeopathy, Flower Essences, Reiki, acupuncture, etc.

Exclusion Criteria:

* Not meet the assumptions of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Self-Reporting Questionnaire (SRQ-20) | (8 months) In 3 times: the first one in the first visit, the second one in the third visit and the last one in the sixth visit.
  The Self-Reporting Questionnaire was developed by Harding et al. (1980), from four other instruments used for screening for possible mental disorders. The development of this instrument was coordinated by World Health Organization (WHO) and aimed to reach a possible instrument to identify cases in primary care services and community, especially in developing countries with lack of services and professionals. The intention of the WHO was to identify cases from the instrument and to encourage planners to provide services and mental health care to the needy population (WHO, 1994).

SECONDARY OUTCOMES:
Spiritual Index of Well-Being Scale (SIWBS) | (8 months) 3 times after the intervention: the first one in the first visit, the second one in the third visit and the last one in the sixth visit
  This instrument, translated and validated into Portuguese from the Index of Spiritual Well-Being Scale (SIWBS) is a research tool that aims to assess the influence of spiritual values in the spiritual welfare of individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan A Guerrini, PhD, Study Chair — Medical School of São Paulo State University (UNESP); Ruth Turrini, PhD, Study Chair — Nursing School of University of São Paulo - (EEUSP)
Locations (1):
- University of Vale do Paraíba, São José dos Campos, São Paulo, Brazil